CLINICAL TRIAL: NCT04313673
Title: Can the Measurement of Transabdominal Cervical Length Predict Preterm Labor During Routine Antenatal Screening Between Weeks 18-22 ?
Brief Title: Transabdominal Cervical Length Predict Preterm Labor During Routine Antenatal Screening
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, erhan hüseyin cömert, physician, Karadeniz Technical University
Other Study IDs: GOLEdvlt
Record Dates: First submitted 2020-03-15; First posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Preterm Labor
Keywords: ultrasonography; transvaginal; transabdominal; second trimester; preterm labor; predict
MeSH Terms: conditions — Obstetric Labor, Premature

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- randomized: Patients who were followed up in our clinic with a diagnosis of preterm labor that spontaneously took action and were born before 37 weeks of gestation will form a group.
  Interventions: Diagnostic Test: second trimester ultrasonography

INTERVENTIONS:
Diagnostic Test: second trimester ultrasonography — Patients undergoing routine antenatal screening between 18-24 weeks and measuring cervical length with transabdominal ultrasonography in the same session

SUMMARY:
Sonographically, cervical length measurement is widely used in obstetrics. Studies have revealed that early detection of short cervix can be a predictor of predicting preterm labor. Transvaginal ultrasonography has been shown as a reference method for the recognition of the short cervix, as well as it may be useful in the transabdominal evaluation in the studies conducted. In addition to the advantages of transvaginal evaluation, it is time consuming and disadvantages of some women during anxiety and discomfort during this procedure. Transabdominal ultrasonography, which provides a non-invasive evaluation, is more preferred by some patients than transvaginal. The aim of this study is to investigate the value of the cervical length measured by transabdominal route, which is a more acceptable method for pregnant women, in predicting preterm birth.

DETAILED DESCRIPTION:
Births that occur before 37th gestational week are an important cause of perinatal morbidity and mortality. Preterm birth accounts for about 12% of all births. Early screening and correct management of pregnant women at risk of preterm birth is essential in reducing perinatal mortality and morbidity associated with prematurity. But the precise prediction and prevention of preterm birth is still an important research topic.

Transabdominal ultrasonography, which provides a non-invasive evaluation, is more preferred by some patients than transvaginal.The aim of this study was to investigate the value of the cervical length measured by transabdominal route, which is a more acceptable method for pregnant women, in predicting preterm birth.

ELIGIBILITY:
Inclusion Criteria:

-Pregnant women who gave birth in our clinic and have a 2nd trimester cervical length measurement

Exclusion Criteria:

* uterin anomaly
* multiple pregnancy cases with a history of cervical surgery
* termination of pregnancy due to fetal or maternal reasons

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — on pregnant women
Study Population: 200 randomized
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-03-10 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
preterm labor | 2 year
  cases were classified as preterm and term

CONTACTS AND LOCATIONS:
Overall Officials: suleyman guven, professor, Study Chair — karadeniz thecnical universty
Locations (1):
- Karadeniz Technical Universty Medical School, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No